CLINICAL TRIAL: NCT05398588
Title: Comparison of Spencer's Muscle Energy Technique and Cyriax Deep Friction Massage on Adhesive Capsulitis
Brief Title: Spencer's Muscle Energy Technique and Cyriax Deep Friction Massage on Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/10257 Huda Ahmed
Record Dates: First submitted 2022-04-21; First posted 2022-06-01 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Adhesive Capsulitis
Keywords: Spencer muscle technique; Cyriax deep friction massage; SHOULDER PAIN
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyriax Deep Friction Massage (Experimental): Cyriax Deep Friction Massage on targeted muscles (Supraspinatus, Infraspinatus, subscapularis, Deltoid and Pectoralis) 3 minutes each muscle (15 mins in total ) x 1 set , 3 days / week
  Interventions: Other: Cyriax Deep Friction Massage
- Spencer Muscle energy technique (Experimental): The Spencer technique will be applied in Abduction, External rotation and Internal rotation for targeting muscles Supraspinatus, Infraspinatus, subscapularis, Deltoid and Pectoralis.
  10 repetitions x 3set , 3 days/weeK
  Interventions: Other: Spencer Muscle energy technique

INTERVENTIONS:
Other: Cyriax Deep Friction Massage — Hotpack : 10 min TENS : 20 min, High frequency(100 Hz pulse ), 3 days/week Kaltenborn mobilization: End range - Anterior, posterior and caudal glides :10 repetitions with 10 sec hold x 3 sets, 3 days/week Cyriax DFM on targeted muscles (Supraspinatus, Infraspinatus, subscapularis, Deltoid and Pectoralis) 3 minutes each muscle (15 mins in total ) x 1 set , 3 days / week
  Arms: Cyriax Deep Friction Massage
Other: Spencer Muscle energy technique — Hotpack : 10 min TENS : 20 min, High frequency(100 Hz pulse ), 3 days/week Kaltenborn mobilization: End range - Anterior, posterior and caudal glides :10 repetitions with 10 sec hold x 3 sets, 3 days/week The Spencer technique will be applied in Abduction, External rotation and Internal rotation for targeting muscles Supraspinatus, Infraspinatus, subscapularis, Deltoid and Pectoralis.
  10 repetitions x 3set , 3 days/week.
  Arms: Spencer Muscle energy technique

SUMMARY:
To compare the effects of Spencer technique and Cyriax deep friction massage on pain, range of motion (ROM) and functional disability of the shoulder in Adhesive capsulitis

DETAILED DESCRIPTION:
Adhesive capsulitis is a common condition of the shoulder characterized by severe pain, stiffness and gradual loss of both active and passive range of motion (ROM) due to progressive fibrosis and contracture of the glenohumeral joint capsule.As a result, capsule gets tighten and shoulder movement restriction happens in a capsular pattern Shoulder external rotation ROM is restricted first followed by shoulder abduction and internal rotation.

The stiffness of the shoulder capsule develops muscle spasm. On assessment one will find tenderness on anterior and lateral gleno-humeral joint line followed by muscle spasm and trigger points in pectoral muscles, scapular muscles and deltoid causing pain over the shoulder girdle.According to Travell and Simons study which is also taken as a reference by M.V.Arjun (2021) stated that AC is a muscular dysfunction model.

It is usually classified into two types. One is primary and other is secondary. The idiopathic cause in which no finding in history or examination explains the reason for onset is known as "Primary Adhesive capsulitis". The disorder develops from a known cause called "Secondary Adhesive capsulitis" According to a study of 2020 by Akshay Date and Luthfur Rahman there are four stages of Adhesive capsulitis. Stage 1 (less than 3 months) is a "painful stage" with moderate pain and reduced movement due to hypertrophic synovitis with hyper vascularity. Stage 2 (3-9 months) is the "Freezing stage" with severe pain and limited shoulder movement due to perivascular synovitis and disorganized collagen deposition and scarring. Stage 3 (10-14 months) is the "Frozen stage" with marked stiffness due to dense and hyper cellular collagenous tissue of the capsule. The last stage 4 (14-24 months) is the "Thawing stage" with minimal pain and gradual improvement in movement.

Although pain and decreased range of motion cause functional limitation of the shoulder but with appropriate treatment and rehabilitation intervention, the severity of disability due to FS is markedly reduced in patients. Physical therapy is often considered the 1st line of treatment option for FS as various exercise and physical therapy modalities help to relieve pain, maintain ROM and restore functions. Out of different manual techniques we will work on Spencer technique and Cyriax deep friction massage and compare their effects.

Spencer muscle energy technique (SMET) is an osteopathic manipulative treatment which is widely used in western practice to treat shoulder problems. It consists of different articulation techniques especially designed to enhance mobility of glenohumeral and scapulothoracic joints by stretching of soft tissue and mobilization of fluid in Adhesive capsulitis patients.To stretch the contracted muscles, ligaments and joint capsules, smooth, rhythmical, passive motion couple with active muscular contraction is required as it includes both active and passive approaches. This procedure required slow stretching of the shoulder joint within the available ROM and maintaining it into the restrictive barrier by a physiotherapist (passive) and creating isometric contraction of muscles against resistance by the patient ( active) followed by a relaxation phase succeeding to the new restrictive barrier. This voluntary isometric contraction of targeted antagonist muscle produces relaxation to agonist muscle and helps reduce the spasms which in turn increase range of which was decreased due to muscle spasm.It also increases blood circulation to the shoulder joint, enhances lymphatic flow and stretches the muscle, ligaments and capsule of the shoulder joint in order to enhance pain-free range of motion.

Different studies such as Anil Rimal (2021), Raksha R et.al (2021) and Mushyyaida (2020) suggested that SMET is effective for reducing pain, increasing ROM and improving functionality in AC.

Another technique used for Adhesive Capsulitis was by James Cyriax, cross-fiber friction massage which is also known as "Deep transverse friction". It is an influential type of soft tissue massage applied transversely to the tissue involved such as ligaments, tendons, muscle bellies, musculotendinous junction and joint capsules.It enhances remodeling and hence reorientation of the collagen fibers in a longitudinal manner. It is a passive technique. The method of applying Deep friction massage on the shoulder is to place the thumb or finger on the shoulder joint line, supraspinatus, subscapularis, Deltoid and pectoralis major and compress. Then move the patient's skin back and forth over the treated fibers perpendicular to the tissue fibers.This will produce transverse movement of collagen fibers that helps in preventing adhesion formation and relaxing muscles. This technique also provides analgesic effects via gate control theory.

There are few studies in literature which prove the effectiveness of Spencer MET and Cyriax DFM on Adhesive Capsulitis. However, there have been no studies which have compared the effectiveness of both the techniques. The rationale behind our study is to determine the most effective technique among Spencer MET and Cyriax DFM. To find out whether Spencer is more effective for the Adhesive Capsulitis patients regarding pain, range of motion and functional disability,as it contains both active and passive approaches as compared to Cyriax DFM or vice versa.

ELIGIBILITY:
Inclusion Criteria:

Both male and female. Unilateral Adhesive capsulitis Primary / idiopathic patients Clinically diagnosed patients with idiopathic Adhesive Capsulitis of Stage 2 and 3. Age group (40-60 years)

Exclusion Criteria:

History of any trauma

* Un-controlled diabetes
* Rotator cuff tears
* Shoulder girdle fracture/dislocation
* Thoracic outlet syndrome
* Any other injury causing shoulder pain and decreased ROM

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) for Pain | 4 weeks
  Visual analogue scale (VAS): It is used for measuring pain. It consists of a line usually 100 mm in length that shows descriptors '0' which means "no pain" and '10' which means "worst pain/ unbearable pain". The rating is measured from the left edge.

SECONDARY OUTCOMES:
Shoulder pain and disability index (SPADI) | 4 week
  It is a self-administered two dimensional questionnaire that evaluates pain and functional activities. It consists of 5 questions regarding an individual's pain and 8 questions regarding a patient's functional assessment .Each questions is given 10 marks, making 50 marks for pain scale and 80 marks for functional assessment. Item scores for each section are averaged to produce separate subscale scores ranging from 0(best) to 100(worst).
  It will be used 2 times/week for 4 weeks.
Range of Motion | 4 weeks
  Goniometer ; It consists of a stationary arm, a moveable arm and a fulcrum. This instrument will measure the range of motion at the shoulder.
  It will be used 2 times/week for 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- Railway Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No